CLINICAL TRIAL: NCT03556904
Title: FOcal Radiation for Oligometastatic Castration-rEsistant Prostate Cancer (FORCE): A Phase II Randomized Trial
Brief Title: FOcal Radiation for Oligometastatic Castration-rEsistant Prostate Cancer (FORCE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.163; HUM00138918 (Other: University of Michigan)
Record Dates: First submitted 2018-03-16; First posted 2018-06-14 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Drug Therapy; enzalutamide; abiraterone; Docetaxel; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care therapy will be up to the treating medical oncologist and is not the study intervention. Current systemic therapy is most commonly a second generation androgen pathway inhibitor, including enzalutamide or abiraterone, although other standard agents (e.g. docetaxel, cabazitaxel) are allowed. Patients should begin systemic treatment within 3 weeks of randomization. Standard of care systemic therapy may continue in the absence of toxicities or other specific criteria per protocol.
  Interventions: Drug: Hormone therapy or chemotherapy
- Standard of Care + Ablative Radiation (Experimental): Standard of care systemic therapy plus radiation. Radiation will start within 8 weeks of randomization and complete by day 84. Standard of care systemic therapy may continue in the absence of toxicities or other specific criteria per protocol.
  Interventions: Radiation: Ablative Radiation Therapy; Drug: Hormone therapy or chemotherapy

INTERVENTIONS:
Radiation: Ablative Radiation Therapy — Radiotherapy will typically be delivered to a total EQD2 (Equivalent dose in 2Gy fractions) that ranges between conventional 30 Gy in 10 fractions, to SBRT (Stereotactic Body Radiation Therapy) with 50 Gy in 5 fractions.
  Arms: Standard of Care + Ablative Radiation
Drug: Hormone therapy or chemotherapy — Current standard of care dosing with standard agents; hormone therapy or chemotherapy.
  Other Names: enzalutamide; abiraterone; docetaxel; cabazitaxel

SUMMARY:
This clinical trial will determine whether the addition of radiotherapy to standard of care systemic therapy improves objective progression-free survival compared to systemic therapy alone in patients with oligometastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have biopsy-confirmed adenocarcinoma of the prostate
* Subjects must discontinue any prior systemic therapies (excluding GnRH agonist/antagonists) without PSA withdrawal effects if using first generation anti-androgens. Luteinizing hormone-releasing hormone (LHRH) analogues must be continued if they have not undergone orchiectomy. (Subjects who recently started systemic therapy for metastatic castration-resistant prostate cancer (mCRPC) are eligible to enroll if new therapy was started ≤ 14 days to consent date.)
* Subjects must have progressive metastatic castration-resistant prostate cancer based on at least one of the following criteria while having castrate levels (<50 ng/dL) of testosterone:
* A) PSA progression defined as a 25% increase over baseline value with an increase in the absolute value of at least 2.0 ng/mL that is confirmed by another PSA level with a minimum of a 1-week interval.
* B) Progression of bidimensionally measurable soft tissue or nodal metastasis by CT scan or MRI based on RECIST criteria
* C) Progression of bone disease on bone scan as defined by two new lesions arising
* Subjects must have oligometastatic prostate cancer, defined as between 1 and ≤5 treatment sites that can be treated within a radiotherapy treatment field.
* Subjects must be medically fit to undergo radiotherapy and systemic therapy as determined by the treating physician.
* Age ≥ 18
* ECOG ≤ 2 (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death)
* No prior invasive malignancy in the past 3-years. Exceptions include non-melanomatous skin cancer and in situ cancers of the bladder or head and neck are permissible.
* Subjects must freely sign informed consent to enroll in the study.
* Subjects must use contraception up to 90 days after last drug dose.

Exclusion Criteria:

* Planned systemic therapy with Radium-223 dichloride or sipuleucel-T
* Tumor requiring emergent radiation in view of provider
* Life expectancy estimate of <3 months
* Presence of known parenchymal brain metastasis
* Uncontrolled intercurrent illness
* Inability to undergo radiotherapy, systemic treatment, CTs or bone scans
* Biopsy proven pure small cell or neuroendocrine prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachery Reichert, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Cancer Center, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Started | 9 | 5
Completed | 1 | 0
Not Completed | 8 | 5
Not completed — Disease Progression after treatment started | 3 | 3
Not completed — Sponsor Termination | 2 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 9 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Median Duration of Response
Description: Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. A patient's designated response at any one time is a combination of the assessment of target lesions, non-target lesions, bone lesions and disease symptoms. Progression in this measure is defined as worsened pain or new sites of disease on imaging. Progression by pain due to prostate cancer requires evidence of disease at the site of pain and one or more palliative intervention (opioid therapy for 10 out of 14 consecutive days, radionuclide therapy or radiation therapy). Response and progression definitions used will be a combination of the criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee v1.1 and the Prostate Cancer Working Group 3.
Time Frame: At 12 Months
Population: NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future
Measure: Median (Standard Deviation); unit: months
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
months | NA (NA) — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future | NA (NA) — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future

2. Secondary Outcome: Median Objective Progression Free Survival (PFS) Time
Description: PFS is defined as the duration of time from start of treatment to date of progression or death (whichever is first). Initiation of other prostate directed therapies (excluding bisphosphonates or RANKL inhibitors) is considered to be progression. Reported as Kaplan-Meier estimates, including median at 12 months and 24 month.
Time Frame: At 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
Months | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future | 26 [22 to 100]

3. Secondary Outcome: Median Prostate Specific Antigen (PSA) PFS
Description: The Median PSA PFS is defined as the median duration of time from start of treatment to date that PSA progression is documented or death occurs (whichever is first). PSA progression is defined as a 25% increase over baseline or nadir whichever is lower and an increase in the absolute value of PSA level by 2 ng/ml. Reported as Kaplan-Meier estimates, including median at 12 months and 24 month.
Time Frame: At 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
months | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future

4. Secondary Outcome: Median Radiographic PFS
Description: Radiographic PFS is defined as the duration of time from start of treatment to date that progression is radio-graphically documented or death occurs (whichever is first). Reported as Kaplan-Meier estimates, including median at 12 months and 24 month.
Time Frame: At 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
Months | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future | 26 [22 to 100]

5. Secondary Outcome: Overall Survival Time
Description: Overall survival (OS) is defined as the duration of time from start of treatment to death. Reported as Kaplan-Meier estimates, including median at 12 months and 24 month.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
months | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future

6. Secondary Outcome: Prostate Cancer Specific Survival Time
Description: Prostate Cancer Specific Survival (PCSS) is defined as the duration of time from start of treatment to death from prostate cancer. Reported as Kaplan-Meier estimates, including median at 12 months and 24 month.
Time Frame: 24 months
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
days | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future

7. Secondary Outcome: Non-irradiated Metastases Free Survival Time
Description: Non-irradiated metastases free survival is defined as the duration of time from start of treatment to the date of progressive disease of a new target lesion, a new non-measurable/non-target lesion or emergence of 2 or more new skeletal lesions on a bone scan. Reported as Kaplan-Meier estimates, including median at 12 months and 24 month.
Time Frame: At 24 months
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
days | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future | NA [NA to NA] — NA- Per biostatistician, values must be reported as NA due to lack of data from insufficient number of participants with events. Data is not available now nor will it be available in the future

8. Secondary Outcome: The Proportion of Patients With Complete PSA Response
Description: The number of patients whose PSA becomes undetectable (≤0.2 ng/ml) will be counted in each treatment arm and divided by the number of patients who received any protocol treatment to provide the proportion of patients with complete PSA response. Complete PSA response is defined as an undetectable PSA (≤0.2 ng/ml).
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
percentage of patients | 67 [30 to 93] | 40 [5 to 85]

9. Secondary Outcome: The Proportion of Patients With a PSA Partial Response 50 (PR50)
Description: The number of patients whose PSA declines by 50% decline (PSA partial response 50 (PR50)) will be counted in each treatment arm and divided by the number of patients who received any protocol treatment to provide the proportion of patients with PR50. PR50 response is defined as a decrease in PSA value by ≥ 50%.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
percentage of patients | 89 [52 to 100] | 60 [15 to 95]

10. Secondary Outcome: The Proportion of Patients With a PSA Partial Response 90 (PR90)
Description: The number of patients whose PSA declines by 90% decline (PSA partial response 90 (PR90)) will be counted in each treatment arm and divided by the number of patients who received any protocol treatment to provide the proportion of patients with PR90. PR90 response is defined as a decrease in PSA value by ≥ 90%.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
percentage of patients | 44 [14 to 79] | 60 [14 to 95]

11. Secondary Outcome: The Proportion of Patients That Respond to Treatment
Description: The measurable disease response rate (CR + PR) will be calculated for patients evaluable for measurable disease response. Complete response (CR) is defined as a disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduced in short axis to <10 mm. There can be no appearance of new lesions. Partial Response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
percentage of patients | 22 [1 to 72] | 20 [5 to 51]

12. Secondary Outcome: Patient-reported Outcome Based on NCCN-FACT FPSI-17 (Version 2)
Description: The National Comprehensive Cancer Network Functional Assessment of Cancer Therapy - Prostate Symptom Index (NFPSI-17), version 2 is used to assess high priority symptoms/QOL concerns in patients with advanced prostate cancer (PC). It is a 17-item survey with a recall period of the past 7 days; scored using a 5 point Likert-type scale. Items are scored from 1-4 with some items reverse scored. Described using means or medians. score range is 0-68 with higher scores indicating better health
Time Frame: measured at 6 and 12 months post starting treatment
Population: score range is 0-68 with higher scores indicating better health
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
Number analyzed (Participants) | 9 | 5
score on a scale
  6 Months | 41.5 [37.5 to 45.4] | 39.1 [33.6 to 44.6]
  12 Months | 41.8 [36.6 to 47.1] | 39.7 [31.0 to 48.4]

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 30 days after the last dose of study treatment; additionally, any serious adverse event occurring more than 30 days after the last study treatment if considered to be related to the study treatment. Data was collected during a 4 year and 7 month period for an average of 20 months per patient.
Arm/Group | Standard of Care | Standard of Care + Ablative Radiation
All-Cause Mortality (participants affected / at risk) | 2/9 | 2/5
Serious Adverse Events (participants affected / at risk) | 3/9 | 0/5
Other Adverse Events (participants affected / at risk) | 9/9 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=9) | Standard of Care + Ablative Radiation (N=5)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Leukemia
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=9) | Standard of Care + Ablative Radiation (N=5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 2 (3) | 1 (1)
Fatigue (General disorders) | 4 (9) | 4 (6)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (4)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 3 (6) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (5)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 2 (6)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain in extremity (General disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) — oral thrush
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — lacerations from fall
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (1) — Enlarged cervical LN
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Chronic myeloid leukemia
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — bilateral lower extremity cramping

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03556904/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT03556904/ICF_001.pdf